CLINICAL TRIAL: NCT00340405
Title: Development of a Biologic Specimen Bank for the Study of Early Markers of Lung Cancer Among Tin Miners in Yunnan, China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999920168; OH92-C-0168
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Lung Cancer
Keywords: Blood; Lung Cancer; Occupational Exposure; Radon; Arsenic; Natural History
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tin Miners in China at risk of lung cancer: Tin Miners in China at risk of lung cancer

SUMMARY:
The overall goal of this project is to identify strategies to reduce lung cancer incidence and mortality. Using a high-risk occupational cohort, our specific objectives are 1) to establish a biologic specimen bank and data bank that can be used for the validation and refinement of potential early markers of lung cancer, and 2) to establish a cohort for the study of environmental (including dietary) and genetic risk factors for lung cancer.

Lung cancer is the leading cause of death from malignant neoplasms in the United States and in many countries around the world. Potential strategies to reduce the incidence and mortality of lung cancer include new methods of early detection and identification and alteration of etiologic factors.

The Yunnan Tin Corporation (YTC), located in Yunnan Province in southern China, is a large, nonferrous-metals industry, formed in 1883 and nationalized after the establishment of the People's Republic in 1949. It is involved principally in the production of tin from the mines around the city of Gejiu. The tin miners at YTC have extremely high rates of lung cancer. Among those at high risk, defined as miners 40+ years old with 10+ years of underground mining and/or smelting experience, more than one percent per year develop lung cancer. These extraordinary lung cancer rates result from combined exposure to radon, arsenic, and tobacco smoking in the form of cigarettes and/or bamboo water pipe.

The study population for the development of a biologic specimen bank for the study of early markers of lung cancer is all YTC miners considered to be at high risk for lung cancer based on their occupation exposure (40+ years old with 10+ years of underground or smelting experience). Currently numbering over 7,000, this high-risk group has been the target for the annual lung cancer screening program at the YTC for the past 20+ years. For each high-risk miner, sputum samples are collected annually, read for cytologic interpretation, and stored in Saccomanno's solution for future early marker research. Screening chest x-rays are also obtained. Subjects are followed annually to determine if any have developed lung cancer. Diagnostic workup of suspicious cases includes an additional sputum sample and histology specimen(s), which are used for diagnostic purposes and also retained for future research.

Additional biologic specimens have also been obtained on screenees for etiologic research, including a one-time collection of whole blood, urine, and toenail clippings. Finger stick bloods and buccal smears for DNA will also be sought....

DETAILED DESCRIPTION:
The overall goal of this project is to identify strategies to reduce lung cancer incidence and mortality. Using a high-risk occupational cohort, our specific objectives are 1) to establish a biologic specimen bank and data bank that can be used for the validation and refinement of potential early markers of lung cancer, and 2) to establish a cohort for the study of environmental (including dietary) and genetic risk factors for lung cancer.

Lung cancer is the leading cause of death from malignant neoplasms in the United States and in many countries around the world. Potential strategies to reduce the incidence and mortality of lung cancer include new methods of early detection and identification and alteration of etiologic factors.

The Yunnan Tin Corporation (YTC), located in Yunnan Province in southern China, is a large, nonferrous-metals industry, formed in 1883 and nationalized after the establishment of the People's Republic in 1949. It is involved principally in the production of tin from the mines around the city of Gejiu. The tin miners at YTC have extremely high rates of lung cancer. Among those at high risk, defined as miners 40+ years old with 10+ years of underground mining and/or smelting experience, more than one percent per year develop lung cancer. These extraordinary lung cancer rates result from combined exposure to radon, arsenic, and tobacco smoking in the form of cigarettes and/or bamboo water pipe.

The study population for the development of a biologic specimen bank for the study of early markers of lung cancer is all YTC miners considered to be at high risk for lung cancer based on their occupation exposure (40+ years old with 10+ years of underground or smelting experience). Currently numbering over 7,000, this high-risk group has been the target for the annual lung cancer screening program at the YTC for the past 20+ years. For each high-risk miner, sputum samples are collected annually, read for cytologic interpretation, and stored in Saccomanno's solution for future early marker research. Screening chest x-rays are also obtained. Subjects are followed annually to determine if any have developed lung cancer. Diagnostic workup of suspicious cases includes an additional sputum sample and histology specimen(s), which are used for diagnostic purposes and also retained for future research.

Additional biologic specimens have also been obtained on screenees for etiologic research, including a one-time collection of whole blood, urine, and toenail clippings. Finger stick bloods and buccal smears for DNA will also be sought.

ELIGIBILITY:
* INCLUSION CRITERIA:

Study participants will be taken from those participating in the annual lung cancer screening examinations conducted by the Labor Protection Institute of the YTC.

Current or retired workers between the ages of 40 and 74.

A history of 10 or more years of underground mining and/or smelting experience.

No proven, active malignancy or serious illness that would interfere with sputum specimen collection.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Yunnan Tin Corporation (YTC), located in Yunnan Province in southern China, is a large, nonferrousmetals industry, formed in 1883 and nationalized after the establishment of the People's Republic in 1949. It is involved principally in the production of tin from the mines around the city of Gejiu. The tin miners at YTC have extremely high rates of lung cancer. Among those at high risk, defined as miners 40+ years old with 10+ years of underground mining and/or smelting experience, more than one percent per year develop lung cancer. These extraordinary lung cancer rates result from combined exposure to radon, arsenic, and tobacco smoking in the form of cigarettes and/or bamboo water pipe. The study population for the development of a biologic specimen bank for the study of early markers of lung cancer@@@is all YTC miners considered to be at high risk for lung cancer based on their occupation exposure (40+ years old with 10+ years of underground or smelting experience).
Sampling Method: Non-Probability Sample
Enrollment: 9759 (Actual)
Dates: Start 1992-04-30 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Identification, validation and refinement of potential early markers of lung cancer | 12/31/2040
  Examining sputum microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Cancer Institute of the Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Qiao YL, Taylor PR, Yao SX, Erozan YS, Luo XC, Barrett MJ, Yan QY, Giffen CA, Huang SQ, Maher MM, Forman MR, Tockman MS. Risk factors and early detection of lung cancer in a cohort of Chinese tin miners. Ann Epidemiol. 1997 Nov;7(8):533-41. doi: 10.1016/s1047-2797(97)00115-4. PMID 9408549
- [Background] Qiao YL, Tockman MS, Li L, Erozan YS, Yao SX, Barrett MJ, Zhou WH, Giffen CA, Luo XC, Taylor PR. A case-cohort study of an early biomarker of lung cancer in a screening cohort of Yunnan tin miners in China. Cancer Epidemiol Biomarkers Prev. 1997 Nov;6(11):893-900. PMID 9367062
- [Background] Taylor PR, Qiao YL, Schatzkin A, Yao SX, Lubin J, Mao BL, Rao JY, McAdams M, Xuan XZ, Li JY. Relation of arsenic exposure to lung cancer among tin miners in Yunnan Province, China. Br J Ind Med. 1989 Dec;46(12):881-6. doi: 10.1136/oem.46.12.881. PMID 2611163
- [Derived] Fan YG, Hu P, Jiang Y, Chang RS, Yao SX, Wang W, He J, Prorok P, Qiao YL. Association between sputum atypia and lung cancer risk in an occupational cohort in Yunnan, China. Chest. 2009 Mar;135(3):778-785. doi: 10.1378/chest.08-1469. PMID 19265088